CLINICAL TRIAL: NCT06998992
Title: Assessing the Reliability of Self-Reported Hepatitis B Vaccination Status in Outpatients: Evaluation of Individuals Born in France and Consulting at the CeGIDD in Saint-Denis.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0006_SMIT
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B; Vaccination; Health Knowledge, Attitudes, Practice; Serologic Tests; Ambulatory Care; Public Health
MeSH Terms: conditions — Hepatitis B; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to find out whether people accurately know their hepatitis B vaccination status. It focuses on individuals born in France who visit a sexual health clinic (CeGIDD) in Saint-Denis. During the consultation, each person is asked whether they think they are vaccinated against hepatitis B. Then, a blood test is done to check if they really are. The goal is to see how often people's answers match their actual medical status. The study also looks at factors like age, gender, education level, and whether they have a regular doctor to understand who is more likely to be unsure or mistaken about their vaccination status. About 200 participants are expected to take part.

ELIGIBILITY:
Inclusion Criteria:

* Patients born in France.
* Consulting at the CeGIDD of Delafontaine Hospital in Saint-Denis.
* Requiring a hepatitis B serology test.

Exclusion Criteria:

- Patients with a history of past hepatitis B infection.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be adults born in France who attend the CeGIDD (sexual health clinic) at Delafontaine Hospital in Saint-Denis. These individuals are seeking care and require a hepatitis B serology test. The population includes people with diverse backgrounds in terms of age, sex, sexual orientation, and education level. Patients with a known history of past hepatitis B infection will be excluded. The study focuses on evaluating the reliability of their self-reported hepatitis B vaccination status compared to serological test results.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who declared being vaccinated against hepatitis B and who are confirmed to be truly vaccinated by serology. | July 2020 - October 2020

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France